CLINICAL TRIAL: NCT00640744
Title: Phase 3 Study of Atorvastatin Effects on Carotid Atherosclerosis
Brief Title: Effect of Short Term Atorvastatin Treatment,80mg/Day on Early Regression of Carotid Artery Atherosclerotic Lesions
Acronym: DCAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baylor College of Medicine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Joel D. Morrisett, Ph.D., Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-18077; HL 063090
Record Dates: First submitted 2008-01-02; First posted 2008-03-21 (Estimated); Last update posted 2010-12-07 (Estimated); Status verified 2010-12

CONDITIONS: Atherosclerosis
Keywords: Atherogenesis; Atheroma; Arteriosclerosis
MeSH Terms: conditions — Atherosclerosis; Plaque, Atherosclerotic; Arteriosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): An untreated carotid plaque will be obtained at the first endarterectomy. Atorvastatin 80mg will be administered for 3 months. The contralateral (treated) plaque will be obtained at the second endarterectomy. Hence, each patient will be his/her own control
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Atorvastatin 80 mg tablet/day for 3 months

SUMMARY:
Atherosclerosis is a disease in which the blood vessels become blocked by plaques (consisting of fat, calcification, and fibrous tissue), reducing blood flow to vital organs and tissues.Blockage of the carotid arteries in the neck is a major cause of stroke. One way of treating carotid atherosclerosis is with cholesterol-lowering drugs called statins. Statins have been shown to reduce the risk of coronary heart disease by 24-40% and risk pf stroke by 11-30%.The purpose of this study is to determine if short term treatment with atorvastatin causes early favorable changes in the plaques that block blood flow through the carotid arteries. These changes can be assessed 1) by taking pictures of the carotid arteries with MRI and Ultrasound before and after statin treatment, and 2) by special studies of the plaques removed from the carotid arteries by surgery.

DETAILED DESCRIPTION:
Candidates for bilateral carotid endarterectomy (CEA) who meet study criteria will provide informed consent before their randomization. Before the first CEA, the patient will have MRI, US, and EBCT exams of both carotids. The most occlusive plaque will be resected at the first CEA. The patient will then receive atorvastatin 80 mg/day for 3 months. Then the second CEA will be performed. Six weeks after the second CEA, the patient will have another MRI, US, and EBCT exam and at 6, 12, and 18 months thereafter. This protocol will allow comparison of the characteristics of the plaque that has been exposed to drug vs the plaque that has not been exposed. It will also allow monitoring the effect of drug on restenosis after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* >18 yrs old
* Expected to have an endarterectomy on each carotid artery
* No contraindications for atorvastatin
* Stable cardiovascular health
* Lipid lowering treatment less than 6 mo duration
* Diabetic included if diabetes is controlled
* Patient is not claustrophobic
* Patient has evaluable carotid plaques.

Exclusion Criteria:

* Patient has had previous carotid endarterectomy,stenting, or other procedure
* Unstable cardiovascular status
* Hypersensitivity to statin therapy
* Neck anatomy preventing acquiring bilateral evaluable plaques
* Weight over 285 lbs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2006-02; Primary Completion 2009-11 (Estimated); Study Completion 2010-02 (Estimated)

PRIMARY OUTCOMES:
Changes in carotid plaque composition as assessed by MRI and histology | 3 months

SECONDARY OUTCOMES:
Changes content of cells, proteins and genes in carotid plaque | 3 months
Changes in content of selected proteins and their encoding genes in carotid plaques | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joel D Morrisett, PhD, Principal Investigator — Baylor College of Medicine; Addison M Taylor, MD, PhD, Study Director — Baylor College of Medicine; William Insull, MD, Study Chair — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Background] Choudhary S, Higgins CL, Chen IY, Reardon M, Lawrie G, Vick GW 3rd, Karmonik C, Via DP, Morrisett JD. Quantitation and localization of matrix metalloproteinases and their inhibitors in human carotid endarterectomy tissues. Arterioscler Thromb Vasc Biol. 2006 Oct;26(10):2351-8. doi: 10.1161/01.ATV.0000239461.87113.0b. Epub 2006 Aug 3. PMID 16888239